CLINICAL TRIAL: NCT04329182
Title: Role of Color Doppler Ultrasonography in Evaluation of Active Sacroiliitis in Ankylosing Spondylitis Patients and Its Relation With Disease Activity
Brief Title: Color Doppler Ultrasonography in Evaluation of Active Sacroiliitis in Ankylosing Spondylitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Salah Eldin Hassan Mohamed Elesseily, Principal investigator, Assiut University
Other Study IDs: Color Doppler Ultrasonography
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Active Sacroiliitis in Ankylosing Spondylitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the role of color Doppler ultrasonography (CDUS) in detection of active sacroiliitis in Ankylosing Spondylitis patients using MRI of the sacroiliac joints as a gold standard.

Evaluate the relation of active sacroiliitis detected by color Doppler ultrasonography (CDUS) with disese activity in patients with ankylosing spondylitis

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is the prototype of the spondyloarthropathies as a chronic inflammatory rheumatic disease presenting mainly with inflammation of the axial skeleton, peripheral arthritis, and enthesitis.

Sacroiliitis is an important sign of AS, and it is used to describe unilateral or bilateral involvement of the sacroiliac joint (SIJ) .

Early diagnosis of AS is important, since some changes associated with the disease are irreversible, and early diagnosis can also improve the ultimate clinical outcomes.

X-ray and magnetic resonance imaging (MRI) are frequently used as image tools to investigate sacroiliitis in AS patients. X-ray could show the structural lesion of sacroiliac joints (SIJs), but could not show the lesions in the early stage of disease. MRI can quantify active in¬flammatory lesions of SIJs.

However, MRI is relatively expensive and time-consuming, and its routine use in patient visits during ther¬apy would be difficult. Another factor that limits usage of MRI is that an important proportion of AS patients have prostheses. Therefore, an easier and cheaper method is needed to detect the degree of spinal inflammation.

Ultrasonography (US) is an inexpensive, non-invasive and non-radiating technique, which can be used in daily clinical practice .

Musculoskeletal ultrasonography (US) has gained increasing attention in many areas of rheumatology . In the area of spondyloarthropathy, Doppler US has been used frequently to assess enthesitis . It was demonstrated that signs of active sacroiliitis could be detected by the color Doppler ultrasonograpy (CDUS) method including increased vascularization in the posterior SIJ and a lower resistance index (RI). The RI could be a quantitative indicator of active sacroiliitis.

Treatment options to AS are limited and mainly consist of non-steroidal anti-inflammatory drugs (NSAIDs) and physical therapy .Efficacy of dis¬ease-modifying anti-rheumatic drugs (DMARDs) such as methotrexate is uncertain to AS.

The introduction of biologic drugs for treatment of AS has led to effective treatment of disease symptoms and signs. However, the effect of these costly drugs on structural damage in addition to the clinical findings is not clear .

ELIGIBILITY:
Inclusion Criteria:

* Age of patients (≥18 and ≤65 years old).
* Diagnosed as Ankylosing Spondylitis defined by the modified New York criteria , and classified as axial Spondyloarthritis according to Assessment in SpondyloArthritis International Society classification criteria.

Exclusion Criteria:

* Diseases mimicking as AS such as :

  * Flourosis of spine,
  * Diffuse idiopathic skeletal hyperostosis (DISH)
  * Degenerative spinal diseases (spondylosis deformans)
* Other seronegative spondyloarthropathy :

  * Psoriatic arthritis ,
  * Reactive Arthritis,
  * Enteropathic Arthritis,
  * Undifferentiated spondyloarthropathy.
* Other causes of sacroiliitis:

  * Osteoarthritis
  * Trauma
  * Infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients involved in the study will be recruited from outpatient clinics and inpatients of Rheumatology, Rehabilitation and Physical Medicine Department, Assiut University Hospitals, Faculty of Medicine.
  Diagnosed as Ankylosing Spondylitis defined by the modified New York criteria , and classified as axial Spondyloarthritis according to Assessment in SpondyloArthritis International Society classification criteria
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
color Doppler ultrasonography (CDUS) in detection of active sacroiliitis in Ankylosing Spondylitis patients | two years
  • Evaluate the role of color Doppler ultrasonography (CDUS) in detection of active sacroiliitis in Ankylosing Spondylitis patients using MRI of the sacroiliac joints as a gold standard